CLINICAL TRIAL: NCT05735353
Title: High-Speed Circuit Resistance Training vs. High-Speed Multidirectional Yoga on Changes in Cognition in Healthy Older Adults.
Brief Title: Sleep, Diet, Exercise and Older Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221319
Record Dates: First submitted 2023-01-12; First posted 2023-02-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Change; Cognitive Decline
Keywords: Circuit Resistance Training; Yoga; Cognition
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Speed Circuit Resistance Training Group (Experimental): Participants in this group will receive high-speed circuit resistance training for 12 consecutive weeks.
  Interventions: Behavioral: High-Speed Circuit Resistance Training
- High-Speed Multidirectional Yoga Group (Experimental): Participants in this group will receive high-speed multidirectional yoga for 12 consecutive weeks.
  Interventions: Behavioral: High-Speed Multidirectional Yoga

INTERVENTIONS:
Behavioral: High-Speed Circuit Resistance Training — three times per week; 45 minutes per session; 12-weeks
  Arms: High-Speed Circuit Resistance Training Group
Behavioral: High-Speed Multidirectional Yoga — two times per week; 60 minutes per session; 12-weeks
  Arms: High-Speed Multidirectional Yoga Group

SUMMARY:
To examine the impacts of a cognitive yoga program and circuit resistance training on cognitive and physical performance with nutrition and sleep as modulating factors in healthy, older adults.

ELIGIBILITY:
Inclusion Criteria:

* Montreal Cognitive Assessment > 23
* No memory loss complaints

Exclusion Criteria:

* Uncontrolled cardiovascular or neuromuscular disease that prevents participation in a training program
* Musculoskeletal impairments or injury that may impact exercise participation
* Visual or hearing impairments
* Neurological disease
* Stroke

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in Executive Function | Baseline, 16 weeks
  Changes in executive function composite score measured by the NIH Toolbox Cognition Module

SECONDARY OUTCOMES:
Changes in Nutritional Status | Baseline, 16 weeks.
  Nutritional status will be assessed by the Nutritionist Pro (Axxya Systems, Redmond, WA), a nutrition analysis software that can be used for diet 24 hour recalls. Participants will be asked to recall food intake for one weekday and one weekend day.
Changes in Sleep Quality as measured by the Pittsburg Sleep Quality Index | Baseline, 16 weeks.
  The Pittsburg Sleep Quality Index has seven component scores that are added to yield one global score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No